CLINICAL TRIAL: NCT01640847
Title: Phase II Trial of Phillips MRI-Guided High Intensity Focused Ultrasound (Sonalleve) and Lyso-thermosensitive Liposomal Doxorubicin (ThermoDox) for Palliation of Painful Bone Metastases
Brief Title: MRI Guided High Intensity Focused Ultrasound (HIFU) and ThermoDox for Palliation of Painful Bone Metastases
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Imunon (Industry)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 106-10-201
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Painful Bone Metastases; Breast Carcinoma; Non-small Cell Lung Cancer; Small Cell Lung Cancer; Adenocarcinoma
Keywords: Painful bone metastases; Bone Cancer; Bone Cancer Pain; Patients with
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Adenocarcinoma; Bone Neoplasms

ARMS (2):
- Arm RT: HIFU plus ThermoDox (Experimental): Index lesion has been treated with EBRT and is currently painful, but these subjects have already received their maximum cumulative EBRT dose.
  Interventions: Drug: High Intensity Focused Ultrasound (HIFU) in combination with ThermoDox
- Arm NRT: HIFU plus ThermoDox (Experimental): Subjects have no yet received any radiation to the index lesion.
  Interventions: Drug: High Intensity Focused Ultrasound (HIFU) in combination with ThermoDox

INTERVENTIONS:
Drug: High Intensity Focused Ultrasound (HIFU) in combination with ThermoDox

SUMMARY:
This study will evaluate treatment with High Intensity Focused Ultrasound (HIFU)in combination with ThermoDox (liposomal doxorubicin) is safe and effective in reducing pain for patients with painful bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast carcinoma, non-small cell lung cancer, small cell lung cancer, or adenocarcinoma of the prostate
* Bone metastases index lesion in the ribs, clavicle, scapula, upper extremities, pelvis, or posterior aspects of the lumbar vertebra L3-L5 or sacral S1-S5.
* Patients will have failed at least one prior attempt or will not be eligible for external beam radiation therapy (EBRT)

Exclusion Criteria:

* Greater than 450 mg/m2 of prior free doxorubicin and/or non-heat activated liposomal doxorubicin
* LVEF < 50%
* Significant Cardiac History
* Brain Metastases
* Contraindication for MR imaging (as incompatible implanted metallic device, weight >250 lbs etc) or known intolerance or allergy to MRI contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Rate of complete pain response | 12 months

SECONDARY OUTCOMES:
Adverse Events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Borys, M.D., Study Director — Imunon